CLINICAL TRIAL: NCT01797263
Title: Pain Outcomes Comparing Yoga Versus Structured Exercise (POYSE) Trial
Acronym: POYSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1100-R
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; yoga; exercise; pain
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga (Experimental): A 12-week yoga intervention modified for Veterans with fibromyalgia. Each weekly session will last approximately 75 minutes. The standardized sequence of yoga poses will be introduced to participants and the instructor will tailor them to the participant's needs and abilities. Deep breathing exercises will be taught and emphasized throughout every session. Participants will be encouraged to exercise according to their limits, rather than rigid adherence to posture techniques. The yoga intervention will be tailored to the individual. It will include low intensity, low impact modified poses adapted with pathophysiologic changes of fibromyalgia in mind. Participants will also be given a Playaway(c) device with guided relaxation exercise recorded on it and asked to listen to it three times a week to reinforce the in person yoga session content.
  Interventions: Other: Yoga
- Structured Exercise (Active Comparator): A 12-week group exercise session consisting of a graded aerobic exercise program. The program will start at low intensity with gradual increases in exercise intensity and duration. Each weekly session will last 75 minutes. The fitness instructor will teach participants to use a table-top ergometer at a sub-maximal level, determine baseline fitness, and develop an individualized exercise prescription. The fitness instructor will provide educational tips on exercise and selection of physical activities. Participants will be given a pedometer and heart rate monitor to track their exercise at home. They will also be given an exercise DVD to use at home.
  Interventions: Other: Structured Exercise

INTERVENTIONS:
Other: Yoga — A 12-week yoga intervention modified for Veterans with fibromyalgia. Each weekly session will last approximately 75 minutes. The standardized sequence of yoga poses will be introduced to participants and the instructor will tailor them to the participant's needs and abilities. Deep breathing exercises will be taught and emphasized throughout every session. Participants will be encouraged to exercise according to their limits, rather than rigid adherence to posture techniques. The yoga intervention will be tailored to the individual. It will include low intensity, low impact modified poses adapted with pathophysiologic changes of fibromyalgia in mind. Participants will also be given a Playaway(c) device with guided relaxation exercise recorded on it and asked to listen to it three times a week to reinforce the in person yoga session content.
  Arms: Yoga
Other: Structured Exercise — A 12-week group exercise session consisting of a graded aerobic exercise program. The program will start at low intensity with gradual increases in exercise intensity and duration. Each weekly session will last 75 minutes. The fitness instructor will teach participants to use a table-top ergometer at a sub-maximal level, determine baseline fitness, and develop an individualized exercise prescription. The fitness instructor will provide educational tips on exercise and selection of physical activities. Participants will be given a pedometer and heart rate monitor to track their exercise at home. They will also be given an exercise DVD to use at home.
  Arms: Structured Exercise

SUMMARY:
The Pain Outcomes comparing Yoga versus Structured Exercise (POYSE) Trial is a 2-arm parallel group, randomized clinical trial to compare the effectiveness of a yoga-based intervention (YOGA) with that of a structured exercise program (SEP) for subjects with fibromyalgia. The study aims are: 1) to compare the interventions' (YOGA vs. SEP) effects on overall fibromyalgia severity at 1 month (early response), 3 months (immediate post-intervention) and at 6 and 9 months (sustained effects); 2) to compare the interventions effects on specific fibromyalgia symptoms (pain, sleep, and fatigue), functional impairment, and related outcomes (quality of life, psychological symptoms); and 3) to compare the cost-effectiveness of the interventions.

DETAILED DESCRIPTION:
This study sample will include 306 Veterans with fibromyalgia. Patients will be randomized to one of two treatment arms. The YOGA arm will involve a standardized 12-week, yoga-based intervention. The yoga intervention will consist of three treatment components: 1) in-person group yoga taught by a certified yoga therapist; 2) a relaxation audio recording for home-use; and 3) a DVD recording to reinforce concepts taught during in-person yoga sessions. Patients randomized to the structured exercise program (SEP) arm will participate in a 12-week exercise program delivered in a group/class format and supervised by a fitness instructor. In addition, SEP patients will receive a DVD (for home use) describing the benefits of aerobic exercise for fibromyalgia, a one-on-one consultation session with the fitness instructor, an individualized exercise prescription, and supervised exercise sessions for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Veterans will be eligible if they have:

* Widespread Pain Index (WPI) greater than 7 and Symptom Severity Scale (SS) greater than 5 or WPI 3-6 and SS greater than 9.
* Symptoms have been present at a similar level for at least 3 months
* The subject does not have a disorder that would otherwise explain the pain
* Moderate pain severity (pain severity score greater than 5)
* No changes in fibromyalgia medications for last 4 weeks
* Access to a working telephone

Exclusion Criteria:

Exclusion criteria includes:

* Severe medical conditions in which exercise is contraindicated (such as significant cardiovascular disease, COPD or asthma needing home oxygen, stroke or TIA in last 6 months, cancer (other than skin cancer) and receiving treatment for it
* Active psychosis
* Hospitalized for psychiatric reasons within the last 6 months
* Active suicidal ideation
* Moderate to severe cognitive impairment
* Involvement in ongoing yoga classes or moderately intense exercise program in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Bair, MD MS, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allsop VL, Schmid AA, Miller KK, Slaven JE, Daggy JK, Froman A, Kline M, Sargent C, French DD, Ang D, Van Puymbroeck M, Schalk NL, Bair MJ. The Pain Outcomes Comparing Yoga vs. Structured Exercise (POYSE) Trial in Veterans With Fibromyalgia: Study Design and Methods. Front Pain Res (Lausanne). 2022 Jul 7;3:934689. doi: 10.3389/fpain.2022.934689. eCollection 2022. PMID 35875477

RESULTS

PARTICIPANT FLOW:
Groups:
- Yoga: A 12-week yoga intervention modified for Veterans with fibromyalgia. Each weekly session will last approximately 75 minutes. The standardized sequence of yoga poses will be introduced to participants and the instructor will tailor them to the participant's needs and abilities. Deep breathing exercises will be taught and emphasized throughout every session. Participants will be encouraged to exercise according to their limits, rather than rigid adherence to posture techniques. The yoga intervention will be tailored to the individual. Participants will also be given a Playaway(c) device with guided relaxation exercise recorded on it and asked to listen to it three times a week to reinforce the in person yoga session content.
Period: Overall Study
Arm/Group | Yoga | Structured Exercise
Started (Baseline) | 129 | 127
1 Month | 96 | 87
3 Month | 87 | 84
6 Month | 90 | 85
9 Month | 92 | 87
Completed | 92 | 87
Not Completed | 37 | 40
Not completed — Withdrawal by Subject | 21 | 25
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 15 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga | Structured Exercise | Total
Number analyzed (Participants) | 129 | 127 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.8) | 56.4 (11.0) | 57.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 88 | 88 | 176
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 47 | 94
  White | 68 | 69 | 137
  More than one race | 7 | 7 | 14
  Unknown or Not Reported | 5 | 2 | 7
Marital Status [Count of Participants; unit: Participants]
  Married/unmarried couple | 76 | 66 | 142
  Divorced/separated | 34 | 46 | 80
  Widowed/never married | 19 | 15 | 34
Employment Status [Count of Participants; unit: Participants]
  Employed | 43 | 40 | 83
  Retired | 43 | 38 | 81
  Unable to work | 36 | 33 | 69
  Other | 7 | 16 | 23
Income comfort level [Count of Participants; unit: Participants]
  Comfortable | 60 | 57 | 117
  Just enough | 47 | 46 | 93
  Not enough | 19 | 23 | 42
  Refused to answer/missing | 3 | 1 | 4
Fibromyalgia Impact Questionnaire-Revised Total [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 90. Higher Score = Worse Outcome
  units on a scale | 51.0 (17.4) | 50.1 (17.5) | 50.4 (17.4)
Fibromyalgia Impact Questionnaire-Revised Difficulty subscale [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 20. Higher Score = Worse Outcome
  units on a scale | 12.7 (6.8) | 12.7 (6.5) | 12.7 (6.6)
Fibromyalgia Impact Questionnaire-Revised Impact subscale [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 100. Higher Score = Worse Outcome
  units on a scale | 10.2 (6.1) | 9.8 (5.8) | 10.0 (5.9)
Fibromyalgia Impact Questionnaire Revised Symptoms subscale [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 100. Higher Score = Worse Outcome
  units on a scale | 28.1 (7.4) | 27.7 (8.1) | 27.9 (7.8)
Brief Pain Inventory Pain Severity [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 40. Higher Score = Worse Outcome
  units on a scale | 6.6 (1.6) | 6.8 (1.6) | 6.7 (1.6)
Patient Health Questionnaire-9 (PHQ-9) Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 27. Higher Score = Worse Outcome
  units on a scale | 11.5 (6.2) | 11.4 (6.3) | 11.5 (6.2)
GAD-7 Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — 0 to 21 with higher scores representing more severe anxiety
  units on a scale | 8.0 (5.9) | 7.7 (5.3) | 7.9 (5.6)
PTSD Checklist of symptoms [Mean (Standard Deviation); unit: units on a scale] — Min: 0, Max: 85 with higher scores representing more severity
  units on a scale | 51.5 (15.4) | 52.6 (14.4) | 52.1 (14.9)
SF-12 Physical Score (health-related quality of life) [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 100. Higher Score = Worse Outcome
  units on a scale | 23.3 (13.7) | 24.0 (18.6) | 23.7 (16.2)
SF-12 Mental Score (health-related quality of life) [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 100. Higher Score = Worse Outcome
  units on a scale | 44.9 (9.5) | 43.7 (9.4) | 44.2 (9.5)
Multi-dimensional fatigue inventory [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 100. Higher Score = Worse Outcome
  units on a scale | 60.2 (22.0) | 59.0 (21.9) | 59.6 (21.9)
MOS Sleep Scale - problems index [Mean (Standard Deviation); unit: units on a scale] — Min:0, Max: 100. Higher Score = Worse Outcome
  units on a scale | 47.0 (11.3) | 46.5 (8.9) | 46.8 (10.2)
Pain catastrophizing scale [Mean (Standard Deviation); unit: units on a scale] — Min: 0. Max: 52. Higher Score = Worse Outcome
  units on a scale | 23.3 (13.7) | 24.0 (13.1) | 23.7 (13.4)
Arthritis self-efficacy scale [Mean (Standard Deviation); unit: units on a scale] — Min: 0, Max: 60. Higher score represents improvement
  units on a scale | 33.4 (12.5) | 33.3 (13.2) | 33.3 (12.8)

OUTCOME MEASURES:

1. Primary Outcome: Fibromyalgia Impact Questionnaire Revised (FIQR) Total Score
Description: This measure will be assessed at Baseline, 1, 3, 6 and 9 months. The 3 month is the primary end point and the 6 and 9 month assessments are for sustained effect. Min:0, Max: 90. Higher Score = Worse Outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 87 | 84
units on a scale | 41.5 (19.3) | 42.2 (20.6)

2. Secondary Outcome: Fibromyalgia Impact Questionnaire-Revised Difficulty Subscale
Description: This represents a subscale of the FIQr and measures patient perceived difficulty related to fibromyalgia. Min:0, Max: 20. Higher Score = Worse Outcome.
Time Frame: 3 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 87 | 84
units on a scale | 10.8 (7.2) | 10.5 (6.9)

3. Secondary Outcome: Fibromyalgia Impact Questionnaire-Revised Impact Subscale
Description: This is a subscale of the FIQr and measures the overall impact of fibromyalgia symptoms. Min:0, Max: 100. Higher Score = Worse Outcome.
Time Frame: 3 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 87 | 84
units on a scale | 7.3 (5.7) | 7.9 (6.2)

4. Secondary Outcome: Fibromyalgia Impact Questionnaire Revised Symptoms Subscale
Description: This subscale of the FIQr provides an overall fibromyalgia symptom score. Min:0, Max: 100. Higher Score = Worse Outcome
Time Frame: 3 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 87 | 84
units on a scale | 23.5 (8.9) | 23.8 (9.7)

5. Secondary Outcome: Brief Pain Inventory (BPI) Severity Subscale
Description: is an 11-item, multidimensional pain measurement tool with demonstrated reliability in patients with arthritis as well as other pain conditions. The BPI rates the intensity of pain as well as the interference of pain with mood, physical activity, work, social activity, relations with others, sleep, and enjoyment of life.Min:0, Max: 40. Higher Score = Worse Outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 87 | 84
units on a scale | 5.6 (1.9) | 5.9 (2.3)

6. Secondary Outcome: PHQ-9 for Depression
Description: will be used to assess depression severity. Several studies have validated the PHQ-9 as a diagnostic measure with excellent psychometric properties. Internal consistency has consistently been shown to be high (Cronbach's alpha > 0.80) and test-retest assessment showed the PHQ-9 to be a responsive and reliable measure of depression treatment outcomes. Min:0, Max: 27. Higher Score = Worse Outcome.
Time Frame: 3 Month
Population: A small number of participants opted to not complete this Outcome measure, causing a discrepancy between this module and the flow module.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 85 | 84
units on a scale | 8.6 (6.1) | 9.8 (6.4)

7. Secondary Outcome: GAD-7 Anxiety Scale
Description: This 7-item scale represent a measure of anxiety symptom severity and provides a score from 0 to 21 with higher scores representing more severe anxiety
Time Frame: 3 Month
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 86 | 84
units on a scale | 6.5 (5.7) | 6.6 (5.4)

8. Secondary Outcome: PTSD Checklist of Symptoms
Description: This 17-item scale assess PTSD symptom severity and provides a severity score; with higher scores representing more severe PTSD. Min: 0, Max: 85 with higher scores representing more severity.
Time Frame: 3 Month
Population: This measure was completed in those participants who screened "positive" for PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 42 | 46
units on a scale | 48.3 (14.7) | 49.0 (17.4)

9. Secondary Outcome: SF-12 Physical Score (Health-related Quality of Life)
Description: The SF-12 is a well-validate measure of health-related quality of life; providing a physical and mental health component summary score. Min:0, Max: 100. Higher Score = Worse Outcome.
Time Frame: 3 Month
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 86 | 84
units on a scale | 17.8 (12.7) | 18.6 (13.9)

10. Secondary Outcome: SF-12 Mental Score (Health-related Quality of Life)
Description: as for outcome 9
Time Frame: 3 Month
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 86 | 84
units on a scale | 46.4 (8.8) | 46.4 (10.0)

11. Secondary Outcome: Multi-dimensional Fatigue Inventory
Description: This scale assesses overall fatigue and has been well-validated and used in other fibromyalgia trials. Min:0, Max: 100. Higher Score = Worse Outcome.
Time Frame: 3 Month
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 85 | 84
units on a scale | 49.2 (24.6) | 51.4 (26.3)

12. Secondary Outcome: MOS Sleep Scale - Problems Index
Description: This scale assesses different aspects of sleep quality and provides an overall index with higher scores representing more severe sleep problems. Min:0, Max: 100. Higher Score = Worse Outcome.
Time Frame: 3 Month
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 86 | 84
units on a scale | 48.5 (10.4) | 44.8 (9.6)

13. Secondary Outcome: Pain Catastrophizing Scale
Description: This 13-item scale assesses pain catastrophizing which has been found to be a predictor of poor treatment response. Min: 0. Max: 52. Higher Score = Worse Outcome.
Time Frame: 3 Month
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 86 | 84
units on a scale | 17.8 (12.7) | 18.6 (13.9)

14. Secondary Outcome: Arthritis Self-efficacy Scale
Description: This scale has been well-validated to assess self-efficacy or confidence in a person's ability to complete a task. Min: 0, Max: 60. Higher score represents improvement.
Time Frame: 3 Month
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Structured Exercise
Number analyzed (Participants) | 86 | 84
units on a scale | 37.2 (12.2) | 37.0 (14.4)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Yoga | Structured Exercise
All-Cause Mortality (participants affected / at risk) | 1/129 | 0/127
Serious Adverse Events (participants affected / at risk) | 2/129 | 4/127
Other Adverse Events (participants affected / at risk) | 26/129 | 29/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga (N=129) | Structured Exercise (N=127)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — Suffered a stroke requiring hospitalization and treatment
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga (N=129) | Structured Exercise (N=127)
Thoughts of self-harm (Psychiatric disorders) | 26 (35) | 29 (46)

LIMITATIONS AND CAVEATS:
Higher than expected study withdrawal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT01797263/Prot_SAP_000.pdf